CLINICAL TRIAL: NCT01433991
Title: An Open-Label, Multicenter Phase 1b/2 Study of E7050 in Combination With E7080 in Subjects With Advanced Solid Tumors (Dose Escalation) and in Subjects With Recurrent Glioblastoma or Unresectable Stage III or Stage IV Melanoma After Prior Systemic Therapy (Expansion Cohort and Phase 2)
Brief Title: A Study of E7050 in Combination With E7080 in Participants With Advanced Solid Tumors (Dose Escalation) and in Participants With Recurrent Glioblastoma or Unresectable Stage III or Stage IV Melanoma After Prior Systemic Therapy (Expansion Cohort and Phase 2)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study was terminated by the sponsor early at the end of Phase 1b due to a change in corporate strategy.
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7050-G000-901
Record Dates: First submitted 2011-09-07; First posted 2011-09-14 (Estimated); Results first posted 2021-06-08 (Actual); Last update posted 2021-06-08 (Actual); Status verified 2021-05

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — N-(2-fluoro-4-((2-(4-(4-methylpiperazin-1-yl)piperidin-1-yl)carbonylaminopyridin-4-yl)oxy)phenyl)-N'-(4-fluorophenyl)cyclopropane-1,1-dicarboxamide; lenvatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1B (Experimental): Participants with unresectable advanced or metastatic solid tumors will receive E7050 in combination with lenvatinib to identify a Maximum Tolerated Dose. Dose escalation will begin at low doses of both E7050 and lenvatinib, and then gradually increase in future cohorts until a recommended combination dose is identified. A dose of E7050 and lenvatinib to be used in combination in Phase 2 will be recommended (RP2 dose). Participants will continue on treatment until disease progression, development of unacceptable toxicity, or withdrawal of consent.
  Interventions: Drug: Golvatinib; Drug: Lenvatinib
- Phase 2 Cohort 1 Arm A: (Experimental): Participants with recurrent glioblastoma (bevacizumab-naïve) will receive E7050 and lenvatinib at the RP2 dose.
  Interventions: Drug: Golvatinib; Drug: Lenvatinib
- Phase 2 Cohort 1 Arm B: (Experimental): Participants with recurrent glioblastoma (bevacizumab-naïve) will receive single agent lenvatinib 24 mg/day (1*4 mg capsule + 2*10 mg capsule) and at time of progression, E7050 add-on therapy at the RP2 dose (in combination with lenvatinib at dose of either the RP2 dose or the most recent dose of single agent lenvatinib, whichever is the lowest).
  Interventions: Drug: Golvatinib; Drug: Lenvatinib
- Phase 2 Cohort 2 Arm C: (Experimental): Participants with unresectable Stage III or Stage IV melanoma and disease progression after prior systemic treatment will receive E7050 and lenvatinib at the RP2 dose.
  Interventions: Drug: Golvatinib; Drug: Lenvatinib
- Phase 2 Cohort 2 Arm D: (Experimental): Participants with unresectable Stage III or Stage IV melanoma and disease progression after prior systemic treatment will receive single agent E7050 400 mg/day.
  Interventions: Drug: Golvatinib

INTERVENTIONS:
Drug: Golvatinib — Participants will receive E7050 50 mg and/or 100 mg tablets. E7050 will be administered orally once daily, in 28-day cycles.
  Other Names: E7050
Drug: Lenvatinib — Participants will receive lenvatinib 1 mg and/or 4 mg and/or 10 mg capsules. Lenvatinib will be administered orally once daily, in 28-day cycles.
  Other Names: E7080
  Arms: Phase 1B; Phase 2 Cohort 1 Arm A:; Phase 2 Cohort 2 Arm C:
Drug: Lenvatinib — Participants will receive lenvatinib 24 mg (1*4 mg capsule + 2*10 mg capsule) capsules. Lenvatinib will be administered orally once daily, in 28-day cycles.
  Other Names: E7080
  Arms: Phase 2 Cohort 1 Arm B:

SUMMARY:
This is a multicenter, open-label, Phase 1b/2 study which will be conducted in two parts: a Phase 1b part comprising a dose escalation and an expansion cohort; and a Phase 2 part which will comprise two cohorts. The purpose of the Phase 1b part is to identify the maximum tolerated dose (MTD) of E7050 and E7080 (lenvatinib) in combination in participants with unresectable advanced or metastatic solid tumors. In the subsequent Phase 1b expansion cohort and Phase 2 cohorts, additional participants with recurrent glioblastoma or unresectable Stage III or Stage IV melanoma and disease progression after prior systemic treatment will be enrolled to confirm the MTD (expansion cohort) and to further explore the clinical activity of E7050 and lenvatinib.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria to be included in this study:

1. Phase 1b: Unresectable advanced or metastatic solid tumors.
2. Phase 1b expansion cohort and Phase 2: Histological confirmed diagnosis of glioblastoma (expansion cohort and Cohort 1) or melanoma (expansion cohort and Cohort 2).

   Phase 1b expansion cohort glioblastoma participants, Phase 2 Cohort 1:
3. No evidence of active central nervous systems (CNS) hemorrhage on baseline scans other than in those participants with recurrent glioblastoma who are stable Grade 1.
4. Participants having first or second recurrence documented by magnetic resonance imaging (MRI), following primary management with surgical resection or biopsy, radiotherapy and up to two prior systemic treatments.
5. If participants is on corticosteroids, they must be on a stable dose for 1 week prior to first dose of study drug.
6. Measurable disease defined as bidimensionally contrast enhancing lesions with clearly defined margins by computerized tomography (CT) or MRI scan, with a minimal diameter of 1 cm, and visible on two axial slices which are preferably at most 5 millimeter (mm) apart with 0 mm skip.

   Phase 1b expansion cohort melanoma participants, Phase 2 Cohort 2:
7. Radiographic/ photographic evidence of disease progression according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) (Appendix 3) after no more than two prior systemic regimens for unresectable Stage III or Stage IV disease.
8. American Joint Committee on Cancer (AJCC) unresectable Stage III or Stage IV melanoma.
9. Measurable disease meeting the following criteria:

   1. At least one lesion of greater than or equal to 1.0 cm in the longest diameter for a non-lymph node or greater than or equal to 1.5 centimeter (cm) in the short-axis diameter for a lymph node which is serially measurable according to RECIST 1.1 using CT/MRI or photography. If there is only one target lesion and it is a non-lymph node, it should have a longest diameter of greater than or equal to 1.5 cm.
   2. Lesions that have had external beam radiotherapy or loco-regional therapies such as radio frequency ablation must show evidence of progressive disease based on RECIST 1.1 to be deemed a target lesion.

   All participants:
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
11. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP less than or equal to 150/90 millimeter of mercury (mmHg) at screening and no change in antihypertensive medications within 1 week before the Screening Visit.
12. Adequate renal function as evidenced by serum creatinine less than or equal to 2.0 milligrams per deciliter (mg/dL) or calculated creatinine clearance greater than or equal to 40 milliliters per minute (mL/min) per the Cockcroft and Gault formula (see Appendix 5).
13. Adequate bone marrow function:

    * Absolute neutrophil count greater than or equal to 1500/mm3 (greater than or equal to 1.5 x 10^3/uL);
    * Platelets greater than or equal to 100,000/mm3 (greater than or equal to 100 x 10^9/L);
    * Hemoglobin greater than or equal to 9.0 g/dL. 14.Adequate blood coagulation function, as evidenced by an International Normalized Ratio (INR) less than or equal to 1.5.
14. Adequate liver function:

    * Bilirubin less than or equal to 1.5 x the upper limit of normal (ULN) except for unconjugated hyperbilirubinemia of Gilbert's syndrome;
    * ALP, ALT, and AST less than or equal to 3 x ULN (less than or equal to 5 x ULN if participant has liver metastases).
15. Males or females age greater than or equal to 18 years at the time of informed consent.
16. All females must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of beta-human chorionic gonadotropin [B-hCG] at the Screening and Baseline Visit (a separate Baseline assessment is not required if a negative Screening pregnancy test was obtained within 72 hours before the first dose of study drug). Females of child-bearing potential, if not practising total abstinence or having a vasectomized partner with confirmed azoospermia, must agree to use two highly effective methods of contraception: e.g., 1) an intrauterine device (IUD) or intrauterine system (IUS); 2) a barrier method such as a condom or occlusive cup (diaphragm or cervical/vault caps) + spermicide (foam, gel, cream, etc.); 3) oral, injected, or implanted hormonal contraceptives throughout the entire study period and for 30 days after study drug discontinuation. Use of a double-barrier method (i.e., use at the same time of a condom + occlusive cup [diaphragm or cervical/vault caps] + spermicide [foam, gel, cream, etc.]) is accepted as two highly effective methods of contraception. The only participants who will be exempt from this requirement are postmenopausal women (defined as women who have been amenorrheic for at least 12 consecutive months, in the appropriate age group, without other known or suspected primary cause) or participants who have been sterilized surgically or who are otherwise proven sterile (i.e., bilateral tubal ligation with surgery at least 1 month prior to dosing, total hysterectomy, or bilateral oophorectomy with surgery at least 1 month prior to dosing). All women who are of reproductive potential and who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 4 weeks prior to dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
17. Male participants who are partners of women of childbearing potential must use a condom + spermicide and their female partners, if of childbearing potential, must use a highly effective method of contraception (see methods described in Inclusion Criterion #18) beginning at least 1 menstrual cycle prior to starting study drug, throughout the entire study period, and for 30 days after the last dose of study drug, unless the male participants are totally abstinent sexually or have undergone a successful vasectomy with confirmed azoospermia or unless the female partners have been sterilized surgically or are otherwise proven sterile (see Inclusion Criterion #16).
18. Voluntary agreement to provide written informed consent and the willingness and ability to comply with all aspects of the protocol.

Exclusion Criteria:

Participants who meet any of the following criteria will be excluded from this study:

1. Phase 1b Dose Escalation: Participants who discontinued prior TK inhibitor (including VEGFR and c-Met receptor targeted therapy) due to toxicity will be ineligible.
2. Phase 1b Dose Escalation (3+3 portion) participants with primary CNS tumors
3. Phase 1b Dose Escalation participants, melanoma participants in expansion cohort and Phase 2 Cohort 2: Participants with untreated or unstable metastases to the central nervous system (CNS) are excluded. participants who have completed local therapy and have discontinued the use of steroids for this indication at least 4 weeks prior to commencing treatment and have remained asymptomatic for at least 4 weeks prior to commencing treatment are eligible.
4. Phase 2: Prior exposure to VEGF-targeted treatment or c-Met or hepatocyte growth factor (HGF) targeted treatment.
5. Phase 2: Active malignancy (except for glioblastoma (Cohort 1) or unresectable Stage III or Stage IV melanoma (Cohort 2); or melanoma in situ, basal or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix) within the past 24 months.

   Phase 1b expansion cohort glioblastoma participants and Phase 2 Cohort 1:
6. More than two recurrences of glioblastoma.
7. Prior bevacizumab treatment.
8. Surgical resection of brain tumor within 4 weeks, or prior stereotactic biopsy within 2 weeks of Screening visit.
9. Prior radiotherapy within 12 weeks unless there is a new area of enhancement consistent with recurrent tumor outside of the radiation field (beyond the high dose region or 80% isodose line), or there is biopsy-proven unequivocal viable tumor on histopathology sampling (e.g., "solid" tumor areas (i.e. greater than 70% tumor cell nuclei in areas), high or progressive increase in MIB-1 proliferation index compared to prior biopsy, or evidence for histological progression or increased anaplasia in the tumor).
10. Participants who have received enzyme-inducing anti epileptic agents within 14 days before the first dose of study drug (e.g., carbamazepine, phenytoin, phenobarbital, primidone, or oxcarbazepine).

    Phase 1b expansion cohort participants with melanoma and Phase 2 Cohort 2:
11. More than two prior systemic regimens for unresectable Stage III or Stage IV disease.

    All participants
12. Prior exposure to E7050 or lenvatinib.
13. Melanoma of intraocular origin.
14. participants who have received any anticancer treatment within 21 days (6 weeks for nitrosureas Cohort 1) or any investigational agent within 30 days prior to the first dose of study drug or who have not recovered from any acute toxicity related to previous anticancer treatment.
15. Major surgery within 3 weeks prior to the first dose of study drug.
16. Participants having greater than 1+ proteinuria on urinalysis will undergo 24-hour urine collection for quantitative assessment of proteinuria. Participants with urine protein greater than or equal to 1 g/24-hour will be ineligible.
17. Inability to take oral medication, gastrointestinal malabsorption, gastrointestinal anastomosis, or any other condition that might affect the absorption of E7050 or lenvatinib.
18. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 6 months of the first dose of study drug; or cardiac arrhythmia requiring medical treatment.
19. Prolongation of QTc interval to greater than 480 msec.
20. Bleeding disorder or thrombotic disorder requiring anticoagulant therapy, such as warfarin, or similar agents requiring therapeutic INR monitoring (treatment with low molecular weight heparin [LMWH] is allowed).
21. Active hemoptysis (bright red blood of at least 0.5 teaspoon) within 3 weeks prior to the first dose of study drug.
22. Active infection (any infection requiring antibiotics).
23. Known intolerance or known hypersensitivity to any of the study drugs (or any of the excipients).
24. Any medical or other condition which, in the opinion of the investigator, would preclude participation in a clinical trial.
25. Females who are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-10-13 (Actual); Primary Completion 2015-03-18 (Actual); Study Completion 2017-03-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Massachusetts General Hospital / Dana Farber Cancer Institute, Boston, Massachusetts

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 2 investigative sites in the United States from 13 October 2011 to 01 March 2017.
Pre-assignment Details: A total of 40 participants were screened, of which 10 were screen failures and 30 participants were enrolled in the study. This study was planned to be conducted in 2 parts: Phase 1b part and Phase 2 part. Study was terminated by the sponsor at the end of Phase 1b due to a change in corporate strategy, hence Phase 2 was not carried out. In this study, a single agent run-in period was conducted prior to the administration of combination treatment in treatment phase.
Groups:
- Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg: Participants received lenvatinib 12 milligram (mg) capsules, orally, once on Day -8, followed by golvatinib 200 mg tablets, orally, once on Day -7 in single agent run in period. Eligible participants who completed run-in period were then entered in combination agent treatment period. In combination agent treatment period, participants received lenvatinib 12 mg capsules, orally, once daily in combination with golvatinib 200 mg tablets, orally, once daily in 28-days treatment cycles until disease progression, development of unacceptable toxicity, or withdrawal of consent (up to approximately 88 weeks).
- Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg: Participants received lenvatinib 20 mg capsules, orally, once on Day -8, followed by golvatinib 200 mg tablets, orally, once on Day -7 in single agent run in period. Eligible participants who completed run-in period were then entered in combination agent treatment period. In combination agent treatment period, participants received lenvatinib 20 mg capsules, orally, once daily in combination with golvatinib 200 mg tablets, orally, once daily in 28-days treatment cycles until disease progression, development of unacceptable toxicity, or withdrawal of consent (up to approximately 88 weeks).
- Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg: Participants received lenvatinib 20 mg capsules, orally, once on Day -8, followed by golvatinib 300 mg tablets, orally, once on Day -7 in single agent run in period. Eligible participants who completed run-in period were then entered in combination agent treatment period. In combination agent treatment period, participants received lenvatinib 20 mg capsules, orally, once daily in combination with golvatinib 300 mg tablets, orally, once daily in 28-days treatment cycles until disease progression, development of unacceptable toxicity, or withdrawal of consent (up to approximately 88 weeks).
- Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg: Participants received lenvatinib 20 mg capsules, orally, once on Day -8, followed by golvatinib 400 mg tablets, orally, once on Day -7 in single agent run in period. Eligible participants who completed run-in period were then entered in combination agent treatment period. In combination agent treatment period, participants received lenvatinib 20 mg capsules, orally, once daily in combination with golvatinib 400 mg tablets, orally, once daily in 28-days treatment cycles until disease progression, development of unacceptable toxicity, or withdrawal of consent (up to approximately 88 weeks).
Period: Pretreatment Phase (Single Agent Run-in)
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Started (30 participants enrolled in Pretreatment Phase (single agent run in period) and 28 went on to receive combination treatment in the Treatment Phase and 2 participants were discontinued after receiving only single-agent therapy in the Pretreatment Phase.) | 5 | 3 | 14 | 8
Completed | 3 | 3 | 14 | 8
Not Completed | 2 | 0 | 0 | 0
Not completed — Did not enter into treatment phase | 2 | 0 | 0 | 0
Period: Treatment Phase (Combination Agent)
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Started | 3 | 3 | 14 | 8
Completed | 1 | 2 | 8 | 2
Not Completed | 2 | 1 | 6 | 6
Not completed — Adverse Event | 1 | 0 | 3 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1
Not completed — Participant Choice | 0 | 0 | 0 | 1
Not completed — Clinical progression | 0 | 1 | 2 | 3
Not completed — Progressive disease | 1 | 0 | 0 | 0
Not completed — Terminated by sponsor | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set (combination treatment) included all participants who received at least 1 dose of combination treatment and had at least 1 postbaseline safety evaluation.
Groups:
- Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg: Participants received lenvatinib 12 mg capsules, orally, once on Day -8, followed by golvatinib 200 mg tablets, orally, once on Day -7 in single agent run in period. Eligible participants who completed run-in period were then entered in combination agent treatment period. In combination agent treatment period, participants received lenvatinib 12 mg capsules, orally, once daily in combination with golvatinib 200 mg tablets, orally, once daily in 28-days treatment cycles until disease progression, development of unacceptable toxicity, or withdrawal of consent (up to approximately 88 weeks).
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg | Total
Number analyzed (Participants) | 3 | 3 | 14 | 8 | 28
Age, Continuous [Median (Full Range); unit: years] | 58.0 [36 to 66] | 63.0 [54 to 65] | 64.5 [41 to 75] | 56.5 [34 to 73] | 62.0 [34 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 7 | 4 | 13
  Male | 2 | 2 | 7 | 4 | 15
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 3 | 3 | 12 | 8 | 26
  Asian | 0 | 0 | 1 | 0 | 1
  Other | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Number of Participants Who Experienced Any Dose Limiting Toxicity (DLT)- Combination Treatment
Description: DLT was defined as toxicity related to the combination therapy and was graded according to Common Terminology Criteria for Adverse Events version 4.0 (CTCAE v4.0). Hematological DLTs were Grade 4 neutropenia for greater than or equal to (>=) 7 days or Grade 3 neutropenia with fever (greater than [>] 38.5 degree Celsius (°C) in axilla), Grade 4 thrombocytopenia or Grade 3 thrombocytopenia with bleeding or lasting >7 days and decrease of hemoglobin of Grade 4. Non-hematological DLTS were Grade 3 fatigue, or a 2 point decline in Eastern Cooperative Oncology Group (ECOG) performance status must persist for >7days, Nausea, vomiting or diarrhea must persist at Grade 3 or 4 despite maximal medical therapy, Grade 4 hypertension or Grade 3 hypertension not able to be controlled by medication and any Grade 3 or higher non-hematological laboratory abnormalities that require hospitalization.
Time Frame: Cycle 1 (Cycle length= 28 days)
Population: The safety analysis set (combination treatment) included all participants who received at least 1 dose of combination treatment and had at least 1 postbaseline safety evaluation. Here, overall number analyzed "N" were the participants who were evaluable for the outcome measure.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg: Eligible participants from single agent run-in period, received lenvatinib 12 mg capsules, orally, once daily in combination with golvatinib 200 mg tablets, orally, once daily in 28-days treatment cycles in combination agent treatment period until disease progression, development of unacceptable toxicity, or withdrawal of consent (up to approximately 88 weeks).
- Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg: Eligible participants from single agent run-in period, received lenvatinib 20 mg capsules, orally, once daily in combination with golvatinib 200 mg tablets, orally, once daily in 28-days treatment cycles in combination agent treatment period until disease progression, development of unacceptable toxicity, or withdrawal of consent (up to approximately 88 weeks).
- Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg: Eligible participants from single agent run-in period, received lenvatinib 20 mg capsules, orally, once daily in combination with golvatinib 300 mg tablets, orally, once daily in 28-days treatment cycles in combination agent treatment period until disease progression, development of unacceptable toxicity, or withdrawal of consent (up to approximately 88 weeks).
- Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg: Eligible participants from single agent run-in period, received lenvatinib 20 mg capsules, orally, once daily in combination with golvatinib 400 mg tablets, orally, once daily in 28-days treatment cycles in combination agent treatment period until disease progression, development of unacceptable toxicity, or withdrawal of consent (up to approximately 88 weeks).
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 3 | 3 | 14 | 6
Participants | 0 | 0 | 4 | 2

2. Primary Outcome: Phase 1b: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of Golvatinib in Combination With Lenvatinib
Description: The MTD was defined as the highest dose level at which no more than 1/6 participants experienced a DLTs, with the next higher dose having at least 0 of 3 or 1 of 6 participants experiencing DLTs. MTD was determined by summarizing the number and percentage of participants with DLTs for the first cycle, by study dosing schedule, initial dosing level and overall for the dose escalation part. The RP2D of golvatinib in Combination with lenvatinib was MTD determined by Dose Escalation Committee (DEC) based on safety, PK and clinical data. DLT was defined as toxicity related to the combination therapy and was graded according to CTCAE v4.0.
Time Frame: Cycle 1 (Cycle length= 28 days)
Population: as for baseline characteristics
Measure: Number; unit: milligram per day (mg/day)
Groups:
- All Cohorts: Golvatinib + Lenvatinib: Eligible participants from single agent run-in period, received lenvatinib 12 mg or 20 mg capsules, orally, once daily in combination with golvatinib 200 mg or 300 mg or 400 mg tablets, orally, once daily in 28-days treatment cycles in combination agent treatment period until disease progression, development of unacceptable toxicity, or withdrawal of consent (up to approximately 88 weeks).
Arm/Group | All Cohorts: Golvatinib + Lenvatinib
Number analyzed (Participants) | 28
milligram per day (mg/day)
  MTD | 300.0
  RP2D | 300.0

3. Primary Outcome: Phase 1b: Maximum Tolerated Dose (MTD) and Recommended Phase 2 Dose (RP2D) of Lenvatinib in Combination With Golvatinib
Description: The MTD was defined as the highest dose level at which no more than 1/6 participants experienced a DLTs, with the next higher dose having at least 0 of 3 or 1 of 6 participants experiencing DLTs. MTD was determined by summarizing the number and percentage of participants with DLTs for the first cycle, by study dosing schedule, initial dosing level and overall for the dose escalation part. The RP2D of lenvatinib in Combination with golvatinib was MTD determined by DEC based on safety, PK and clinical data. DLT was defined as toxicity related to the combination therapy and was graded according to CTCAE v4.0.
Time Frame: Cycle 1 (Cycle length= 28 days)
Population: as for baseline characteristics
Measure: Number; unit: mg/day
Groups:
- All Cohorts: Lenvatinib + Golvatinib: Eligible participants from single agent run-in period, received lenvatinib 12 mg or 20 mg capsules, orally, once daily in combination with golvatinib 200 mg or 300 mg or 400 mg tablets, orally, once daily in 28-days treatment cycles in combination agent treatment period until disease progression, development of unacceptable toxicity, or withdrawal of consent (up to approximately 88 weeks).
Arm/Group | All Cohorts: Lenvatinib + Golvatinib
Number analyzed (Participants) | 28
mg/day
  MTD | 20.0
  RP2D | 20.0

4. Secondary Outcome: Phase 1b: Number of Participants With Clinically Significant Change From Baseline in Laboratory Values- Combination Treatment
Time Frame: From baseline up to approximately 5 years 5 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 3 | 3 | 14 | 8
Participants | 0 | 0 | 0 | 0

5. Secondary Outcome: Phase 1b: Number of Participants With Clinically Significant Change From Baseline in Vital Signs Values- Combination Treatment
Time Frame: From baseline up to approximately 5 years 5 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 3 | 3 | 14 | 8
Participants | 0 | 0 | 0 | 0

6. Secondary Outcome: Phase 1b: Number of Participants With Abnormal 12-lead Electrocardiogram (ECG) Values- Combination Treatment
Time Frame: From baseline up to approximately 5 years 5 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 3 | 3 | 14 | 8
Participants
  Baseline and post-baseline data | 3 | 3 | 13 | 8
  At least 1 post-baseline increase of greater than (>) 30 millisecond (msec) | 2 | 0 | 1 | 4
  At least 1 post-baseline increase of > 60 msec | 1 | 0 | 0 | 0
  At least 1 post-baseline value of > 450 msec | 2 | 2 | 8 | 4
  At least 1 post-baseline value of > 480 msec | 1 | 0 | 4 | 1
  At least 1 post-baseline value of > 500 msec | 1 | 0 | 1 | 0

7. Secondary Outcome: Phase 1b: Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)- Combination Treatment
Time Frame: From baseline up to approximately up to 5 years 5 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 3 | 3 | 14 | 8
Participants
  TEAEs | 3 | 3 | 14 | 8
  SAEs | 2 | 1 | 8 | 3

8. Secondary Outcome: Phase 1b: Cmax; Maximum Observed Plasma Concentration for Golvatinib When Administered as a Single Agent at Day -7
Time Frame: Day -7: 0-24 hours post-dose
Population: The pharmacokinetic (PK) analysis set included participants who had at least 1 evaluable plasma concentration.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 5 | 3 | 6 | 8
nanograms per milliliter (ng/mL) | 2160 (848) | 1710 (1410) | 3020 (2130) | 3930 (1800)

9. Secondary Outcome: Phase 1b: Cmax; Maximum Observed Plasma Concentration for Lenvatinib When Administered as a Single Agent at Day -8
Time Frame: Day -8: 0-24 hours post-dose
Population: The PK analysis set included participants who had at least 1 evaluable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 5 | 3 | 6 | 8
ng/mL | 174 (88.0) | 393 (75.0) | 297 (159) | 388 (250)

10. Secondary Outcome: Phase 1b: Tmax; Time to Reach the Maximum Plasma Concentration (Cmax) for Golvatinib When Administered as a Single Agent at Day -7
Time Frame: Day -7: 0-24 hours post-dose
Population: The PK analysis set included participants who had at least 1 evaluable plasma concentration.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 5 | 3 | 6 | 8
hours | 2.00 [1.43 to 11.6] | 4.00 [3.02 to 4.08] | 2.54 [1.95 to 4.08] | 2.54 [1.98 to 7.92]

11. Secondary Outcome: Phase 1b: Tmax; Time to Reach the Maximum Plasma Concentration (Cmax) for Lenvatinib When Administered as a Single Agent at Day -8
Time Frame: Day -8: 0-24 hours post-dose
Population: The PK analysis set included participants who had at least 1 evaluable plasma concentration.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 5 | 3 | 6 | 8
hours | 3.00 [1.00 to 3.08] | 2.00 [2.00 to 2.92] | 3.01 [1.93 to 8.00] | 3.00 [1.00 to 23.50]

12. Secondary Outcome: Phase 1b: AUC24; Area Under the Plasma Concentration-time Curve From Time 0 to Time 24 Hours for Golvatinib When Administered as Single Agent at Day -7
Time Frame: Day -7: 0-24 hours post-dose
Population: The PK analysis set included participants who had at least 1 evaluable plasma concentration. Here, overall number analyzed "N" were the participants who were evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter(ng*h/mL)
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 4 | 3 | 6 | 8
nanogram*hour per milliliter(ng*h/mL) | 25600 (6720) | 19300 (14000) | 34400 (25600) | 50000 (27900)

13. Secondary Outcome: Phase 1b: AUC24; Area Under the Plasma Concentration-time Curve From Time 0 to Time 24 Hours for Lenvatinib When Administered as Single Agent at Day -8
Time Frame: Day -8: 0-24 hours post-dose
Population: The PK analysis set included participants who had at least 1 evaluable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 5 | 3 | 6 | 8
ng*h/mL | 1540 (581) | 2690 (75.7) | 2620 (1160) | 3200 (2210)

14. Secondary Outcome: Phase 1b: AUCt; Area Under the Plasma Concentration-time Curve From Time 0 to Time t Over the Dosing Interval for Golvatinib When Administered as Single Agent at Day -7
Time Frame: Day -7: 0-24 hours post-dose
Population: The PK analysis set included participants who had at least 1 evaluable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 5 | 3 | 6 | 8
ng*h/mL | 26500 (6380) | 34700 (27900) | 38000 (25400) | 64000 (33000)

15. Secondary Outcome: Phase 1b: AUCt; Area Under the Plasma Concentration-time Curve From Time 0 to Time t Over the Dosing Interval for Lenvatinib When Administered as Single Agent at Day -8
Time Frame: Day -8: 0-24 hours post-dose
Population: PK analysis set included participants who had at least 1 evaluable plasma concentration.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 5 | 3 | 6 | 8
ng*h/mL | 1800 (697) | 3030 (254) | 3030 (1260) | 3780 (2630)

16. Secondary Outcome: Phase 1b: AUC∞; Area Under the Plasma Concentration-time Curve From Time 0 to Infinity Calculated Using the Observed Value for the Last Quantifiable Concentration for Golvatinib When Administered as Single Agent at Day -7
Time Frame: Day -7: 0-24 hours post-dose
Population: PK analysis set included participants who had at least 1 evaluable plasma concentration. Here overall number analyzed "N" were the participants who were evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 0 | 2 | 1 | 0
ng*h/mL |  | 58300 (23500) | 51200 (NA) — Standard deviation could not be calculated because only one participant was available for evaluation. |

17. Secondary Outcome: Phase 1b: AUC∞; Area Under the Plasma Concentration-time Curve From Time 0 to Infinity Calculated Using the Observed Value for the Last Quantifiable Concentration for Lenvatinib When Administered as Single Agent at Day -8
Time Frame: Day -8: 0-24 hours post-dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 5 | 3 | 5 | 8
ng*h/mL | 1890 (693) | 3060 (250) | 2930 (1360) | 3910 (2680)

18. Secondary Outcome: Phase 1b: t1/2; Terminal Elimination Half-life for Golvatinib When Administered as Single Agent at Day -7
Time Frame: Day-7: 0-24 hours post-dose
Population: The PK analysis set included participants who had at least 1 evaluable plasma concentration. Here overall number analyzed "N" were the participants who were evaluable for the outcome measure.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 0 | 2 | 1 | 2
hours |  | 34.6 (1.77) | 30.7 (NA) — Standard deviation could not be calculated because only one participant was available for evaluation. | 57.0 (1.70)

19. Secondary Outcome: Phase 1b: t1/2; Terminal Elimination Half-life for Lenvatinib When Administered as Single Agent at Day -8
Time Frame: Day -8: 0-24 hours post-dose
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 5 | 3 | 5 | 8
hours | 11.2 (3.27) | 14.6 (6.69) | 12.0 (5.49) | 14.4 (6.86)

20. Secondary Outcome: Phase 1b: CL/F; Apparent Clearance After Extravascular Administration Calculated Using the Observed Value of the Last Quantifiable Concentration for Golvatinib When Administered as Single Agent at Day -7
Time Frame: Day -7: 0-24 hours post-dose
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 0 | 2 | 1 | 0
liter per hour (L/h) |  | 3.74 (1.51) | 5.87 (NA) — Standard deviation could not be calculated because only one participant was available for evaluation. |

21. Secondary Outcome: Phase 1b: CL/F; Apparent Clearance After Extravascular Administration Calculated Using the Observed Value of the Last Quantifiable Concentration for Lenvatinib When Administered as Single Agent at Day -8
Time Frame: Day -8: 0-24 hours post-dose
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 5 | 3 | 5 | 8
liter per hour (L/h) | 7.01 (2.31) | 6.57 (0.556) | 8.63 (5.33) | 7.23 (4.25)

22. Secondary Outcome: Phase 1b: Vz/F; Apparent Volume of Distribution at Terminal Phase for Golvatinib When Administered as Single Agent at Day -7
Time Frame: Day -7: 0-24 hours post-dose
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: liter (L)
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 0 | 2 | 1 | 0
liter (L) |  | 188 (84.9) | 260 (NA) — Standard deviation could not be calculated because only one participant was available for evaluation. |

23. Secondary Outcome: Phase 1b: Vz/F; Apparent Volume of Distribution at Terminal Phase for Lenvatinib When Administered as Single Agent at Day -8
Time Frame: Day -8: 0-24 hours post dose
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: liter (L)
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 5 | 3 | 5 | 8
liter (L) | 112 (53.4) | 135 (55.1) | 182 (209) | 137 (87.5)

24. Secondary Outcome: Phase 1b: Cmax; Maximum Observed Plasma Concentration for Golvatinib and Lenvatinib When Administered in Combination Treatment as Single Dose on Day 1 Cycle 1
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (cycle length is 28 days)
Population: PK analysis set included participants who had at least 1 evaluable plasma concentration. Here overall number analyzed "N" were the participants who were evaluable for the outcome measure. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 3 | 3 | 6 | 8
ng/mL
  Golvatinib: Cycle 1 Day 1 | 2890 (1080) | 1990 (1470) | 3050 (1030) | 4820 (1510)
  Lenvatinib: Cycle 1 Day 1: number analyzed (Participants) | 3 | 2 | 5 | 7
  Lenvatinib: Cycle 1 Day 1 | 182 (137) | 315 (35.4) | 258 (148) | 251 (144)

25. Secondary Outcome: Phase 1b: Cmax; Maximum Observed Plasma Concentration for Golvatinib and Lenvatinib When Administered in Combination Treatment as Multiple Dose on Day 1 Cycle 2
Time Frame: Cycle 2 Day 1: 0-24 hours post-dose (cycle length is 28 days)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 1 | 2 | 5 | 4
ng/mL
  Golvatinib: Cycle 2 Day 1 | 3540 (NA) — Standard deviation could not be calculated because only one participant was available for evaluation. | 2750 (870) | 3570 (1350) | 6920 (4130)
  Lenvatinib: Cycle 2 Day 1 | 66.3 (NA) — Standard deviation could not be calculated because only one participant was available for evaluation. | 356 (76.4) | 245 (110) | 408 (250)

26. Secondary Outcome: Phase 1b: Tmax; Time to Reach the Maximum Plasma Concentration (Cmax) for Golvatinib and Lenvatinib When Administered in Combination Treatment as Single Dose on Day 1 Cycle 1
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (cycle length is 28 days)
Population: The PK analysis set included participants who had at least 1 evaluable plasma concentration. Here overall number analyzed "N" were the participants who were evaluable for the outcome measure. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given time points.
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 3 | 3 | 6 | 8
hours
  Golvatinib: Cycle 1 Day 1 | 3.02 [2.12 to 4.02] | 4.00 [2.03 to 4.08] | 3.52 [1.98 to 8.05] | 3.00 [0.98 to 4.13]
  Lenvatinib: Cycle 1 Day 1: number analyzed (Participants) | 3 | 2 | 5 | 7
  Lenvatinib: Cycle 1 Day 1 | 3.02 [2.12 to 4.02] | 2.02 [2.00 to 2.03] | 3.95 [1.98 to 4.03] | 3.98 [2.00 to 4.13]

27. Secondary Outcome: Phase 1b: Tmax; Time to Reach the Maximum Plasma Concentration (Cmax) for Golvatinib and Lenvatinib When Administered in Combination Treatment as Multiple Dose on Day 1 Cycle 2
Time Frame: Cycle 2 Day 1: 0-24 hours post-dose (cycle length is 28 days)
Population: as for outcome 16
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 1 | 2 | 5 | 4
hours
  Golvatinib: Cycle 2 Day 1 | 8.05 [8.05 to 8.05] | 2.00 [1.00 to 3.00] | 2.97 [1.02 to 3.97] | 3.53 [3.00 to 7.92]
  Lenvatinib: Cycle 2 Day 1 | 10.55 [10.55 to 10.55] | 3.00 [2.00 to 4.00] | 3.90 [2.03 to 3.97] | 3.53 [2.00 to 7.92]

28. Secondary Outcome: Phase 1b: AUC24; Area Under the Plasma Concentration-time Curve From Time 0 to Time 24 Hours for Golvatinib and Lenvatinib When Administered in Combination Treatment as Single Dose on Day 1 Cycle 1
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (cycle length is 28 days)
Population: as for outcome 24
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 3 | 3 | 6 | 8
ng*h/mL
  Golvatinib: Cycle 1 Day 1 | 33800 (4270) | 22100 (15900) | 38700 (21700) | 60400 (26200)
  Lenvatinib: Cycle 1 Day 1: number analyzed (Participants) | 3 | 2 | 5 | 7
  Lenvatinib: Cycle 1 Day 1 | 1460 (922) | 2370 (35.4) | 2290 (1250) | 2390 (1710)

29. Secondary Outcome: Phase 1b: AUC24; Area Under the Plasma Concentration-time Curve From Time 0 to Time 24 Hours for Golvatinib and Lenvatinib When Administered in Combination Treatment as Multiple Dose on Day 1 Cycle 2
Time Frame: Cycle 2 Day 1: 0-24 hours post-dose (cycle length is 28 days)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 1 | 2 | 5 | 4
ng*h/mL
  Golvatinib: Cycle 2 Day 1 | 68700 (NA) — Standard deviation could not be calculated because only one participant was available for evaluation. | 45000 (29700) | 57100 (25300) | 138000 (98900)
  Lenvatinib: Cycle 2 Day 1 | 1120 (NA) — Standard deviation could not be calculated because only one participant was available for evaluation. | 3060 (247) | 2380 (1430) | 4320 (3860)

30. Secondary Outcome: Phase 1b: AUCt; Area Under the Plasma Concentration-time Curve From Time 0 to Time t Over the Dosing Interval for Golvatinib and Lenvatinib When Administered in Combination Treatment as Single Dose on Day 1 Cycle 1
Time Frame: Cycle 1 Day 1: 0-24 hours post-dose (cycle length is 28 days)
Population: The PK analysis set included participants who had at least 1 evaluable plasma concentration. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given time points.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 5 | 3 | 6 | 8
ng*h/mL
  Golvatinib: Cycle 1 Day 1: number analyzed (Participants) | 3 | 3 | 6 | 8
  Golvatinib: Cycle 1 Day 1 | 34000 (4290) | 22200 (15900) | 39800 (21800) | 60800 (26700)
  Lenvatinib: Cycle 1 Day 1: number analyzed (Participants) | 5 | 2 | 5 | 7
  Lenvatinib: Cycle 1 Day 1 | 1470 (921) | 2370 (42.4) | 2400 (1270) | 2400 (1730)

31. Secondary Outcome: Phase 1b: AUCt; Area Under the Plasma Concentration-time Curve From Time 0 to Time t Over the Dosing Interval for Golvatinib and Lenvatinib When Administered in Combination Treatment as Multiple Dose on Day 1 Cycle 2
Time Frame: Cycle 2 Day 1: 0-24 hours post-dose (cycle length is 28 days)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 1 | 2 | 5 | 4
ng*h/mL
  Golvatinib: Cycle 2 Day 1 | 68700 (NA) — Standard deviation could not be calculated because only one participant was available for evaluation. | 45200 (29500) | 57100 (25300) | 138000 (98700)
  Lenvatinib: Cycle 2 Day 1 | 1120 (NA) — Standard deviation could not be calculated because only one participant was available for evaluation. | 3060 (255) | 2380 (1430) | 4330 (3850)

32. Secondary Outcome: Phase 1b: CLss/F; Apparent Clearance After Extravascular Administration Calculated Using the Observed Value of the Last Quantifiable Concentration for Golvatinib and Lenvatinib When Administered in Combination Treatment as Multiple Dose on Day 1 Cycle 2
Time Frame: Cycle 2 Day 1: 0-24 hours post-dose (cycle length is 28 days)
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: liter per hour (L/h)
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 0 | 2 | 0 | 3
liter per hour (L/h)
  Golvatinib: Cycle 2 Day 1 |  | 5.69 (3.76) |  | 3.49 (1.81)
  Lenvatinib: Cycle 2 Day 1 |  | 6.58 (0.54) |  | 7.96 (5.72)

33. Secondary Outcome: Phase 1b: Rac(AUC); Accumulation Ratio Based on AUC Calculated as AUC24 at Steady State/AUC24 for Golvatinib and Lenvatinib When Administered in Combination Treatment as Multiple Dose on Day 1 Cycle 2
Time Frame: Cycle 2 Day 1: 0-24 hours post-dose (cycle length is 28 days)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 1 | 2 | 5 | 4
ratio
  Golvatinib: Cycle 2 Day 1 | 2.35 (NA) — Standard deviation could not be calculated because only one participant was available for evaluation. | 3.96 (2.14) | 1.90 (0.905) | 2.10 (0.254)
  Lenvatinib: Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 3 | 4
  Lenvatinib: Cycle 2 Day 1 | 1.88 (NA) — Standard deviation could not be calculated because only one participant was available for evaluation. | 1.29 (0.127) | 0.928 (0.295) | 1.61 (0.670)

34. Secondary Outcome: Phase 1b: Rac(Cmax); Accumulation Ratio Based on Cmax Calculated as Cmax at Steady State/Cmax for Golvatinib and Lenvatinib When Administered in Combination Treatment as Multiple Dose on Day 1 Cycle 2
Time Frame: Cycle 2 Day 1: 0-24 hours post-dose (cycle length is 28 days)
Population: as for outcome 26
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 1 | 2 | 5 | 4
ratio
  Golvatinib: Cycle 2 Day 1 | 2.11 (NA) — Standard deviation could not be calculated because only one participant was available for evaluation. | 3.16 (2.24) | 1.30 (0.481) | 1.49 (0.319)
  Lenvatinib: Cycle 2 Day 1: number analyzed (Participants) | 1 | 2 | 3 | 4
  Lenvatinib: Cycle 2 Day 1 | 1.44 (NA) — Standard deviation could not be calculated because only one participant was available for evaluation. | 1.13 (0.120) | 1.17 (0.556) | 1.63 (1.27)

35. Secondary Outcome: Phase 1b: Objective Response Rate (ORR); Combination Treatment
Description: ORR was assessed by the investigator based on Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1. ORR was defined as the percentage of participants with confirmed best overall response (BOR) of complete response (CR) or partial response (PR). CR was defined as the disappearance of all target and non-target lesions (non-lymph nodes). All pathological lymph nodes (whether target or non-target) must have a reduction in their short axis to less than (<)10 millimeters (mm). PR was defined as at least a 30 percent (%) decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: From the date of the first dose of study drug to the date of the first documentation of disease progression or death, whichever occurred first (approximately up to 5 years 5 months)
Population: Safety analysis set (combination treatment) included all participants who received at least 1 dose of combination treatment and had at least 1 postbaseline safety evaluation.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
Number analyzed (Participants) | 3 | 3 | 14 | 8
percentage of participants | 0 [NA to NA] — The 95% confidence interval could not be estimated due to insufficient number of participants with event during the study. | 0 [NA to NA] — The 95% confidence interval could not be estimated due to insufficient number of participants with event during the study. | 28.6 [8.4 to 58.1] | 12.5 [0.3 to 52.7]

ADVERSE EVENTS:
Time Frame: From baseline up to approximately 5 years 5 months
Arm/Group | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 0/14 | 3/8
Serious Adverse Events (participants affected / at risk) | 2/3 | 1/3 | 8/14 | 3/8
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 13/14 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg (N=3) | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg (N=3) | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg (N=14) | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg (N=8)
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Intestinal Perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Device Occlusion (General disorders) | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Lung Infection (Infections and infestations) | 0 | 1 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Bile Duct Obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Electrocardiogram Qt Prolonged (Investigations) | 1 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Urinary tract infection enterococcal (Infections and infestations) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: Lenvatinib 12 mg + Golvatinib 200 mg (N=3) | Cohort 2: Lenvatinib 20 mg + Golvatinib 200 mg (N=3) | Cohort 3: Lenvatinib 20 mg + Golvatinib 300 mg (N=14) | Cohort 4: Lenvatinib 20 mg + Golvatinib 400 mg (N=8)
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 13 | 5
Vomiting (Gastrointestinal disorders) | 3 | 2 | 9 | 6
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 5 | 3
Constipation (Gastrointestinal disorders) | 1 | 0 | 8 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 1 | 3 | 1
Oral Pain (Gastrointestinal disorders) | 0 | 2 | 2 | 0
Abdominal Distension (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Dry Mouth (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Ascites (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Anal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastrointestinal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Glossodynia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Lip Dry (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oesophageal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Tongue Discolouration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Tongue Geographic (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 2 | 3 | 11 | 5
Oedema Peripheral (General disorders) | 1 | 1 | 3 | 1
Chills (General disorders) | 0 | 0 | 4 | 1
Asthenia (General disorders) | 2 | 0 | 1 | 1
Pain (General disorders) | 0 | 0 | 4 | 0
Pyrexia (General disorders) | 0 | 1 | 2 | 0
Influenza Like Illness (General disorders) | 0 | 0 | 1 | 0
Injection Site Nodule (General disorders) | 0 | 0 | 1 | 0
Injection Site Pain (General disorders) | 0 | 0 | 1 | 0
Injection Site Swelling (General disorders) | 0 | 0 | 1 | 0
Malaise (General disorders) | 0 | 1 | 0 | 0
Peripheral Swelling (General disorders) | 0 | 0 | 1 | 0
Suprapubic Pain (General disorders) | 0 | 0 | 1 | 0
Decreased Appetite (Metabolism and nutrition disorders) | 3 | 2 | 10 | 5
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 7 | 4
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 6 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 5 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 3 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 0
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 6 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 4 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 3 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Increased Upper Airway Secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Aspartate Aminotransferase Increased (Investigations) | 1 | 0 | 10 | 3
Blood Alkaline Phosphatase Increased (Investigations) | 0 | 0 | 8 | 1
Lipase Increased (Investigations) | 1 | 0 | 3 | 2
Blood Creatine Phosphokinase Increased (Investigations) | 0 | 0 | 3 | 1
Electrocardiogram Qt Prolonged (Investigations) | 0 | 0 | 2 | 1
Weight Decreased (Investigations) | 0 | 1 | 3 | 0
White Blood Cell Count Decreased (Investigations) | 0 | 0 | 2 | 2
Neutrophil Count Decreased (Investigations) | 0 | 0 | 2 | 1
Platelet Count Decreased (Investigations) | 0 | 0 | 1 | 2
Amylase Increased (Investigations) | 0 | 0 | 3 | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 3 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 1
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 0
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 1
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0
Bone Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Flank Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle Twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Musculoskeletal Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Tendon Discomfort (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Blood Albumin Decreased (Investigations) | 0 | 0 | 1 | 0
Blood Creatinine Increased (Investigations) | 0 | 0 | 1 | 1
Blood Sodium Decreased (Investigations) | 0 | 0 | 1 | 0
Blood Thyroid Stimulating Hormone Decreased (Investigations) | 0 | 0 | 1 | 0
Blood Thyroid Stimulating Hormone Increased (Investigations) | 0 | 0 | 1 | 0
Clostridium Test Positive (Investigations) | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1 | 4 | 2
Dysgeusia (Nervous system disorders) | 0 | 1 | 3 | 1
Headache (Nervous system disorders) | 0 | 0 | 3 | 0
Peripheral Sensory Neuropathy (Nervous system disorders) | 0 | 0 | 0 | 3
Tremor (Nervous system disorders) | 0 | 0 | 3 | 0
Memory Impairment (Nervous system disorders) | 0 | 0 | 2 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0
Mental Impairment (Nervous system disorders) | 1 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 0 | 1 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 1 | 6 | 2
Deep Vein Thrombosis (Vascular disorders) | 0 | 0 | 1 | 0
Hot Flush (Vascular disorders) | 0 | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 0 | 1 | 0
Orthostatic Hypotension (Vascular disorders) | 0 | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 0 | 6 | 1
Pneumonia (Infections and infestations) | 1 | 0 | 1 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 2 | 0
Abdominal Abscess (Infections and infestations) | 0 | 0 | 1 | 0
Bacteriuria (Infections and infestations) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Clostridium Difficile Colitis (Infections and infestations) | 0 | 0 | 1 | 0
Fungal Infection (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Herpes Simplex (Infections and infestations) | 0 | 0 | 1 | 0
Kidney Infection (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1 | 0
Oral Infection (Infections and infestations) | 0 | 1 | 0 | 0
Sinusitis Bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 0 | 0 | 1 | 0
Viral Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 4 | 1
Palmar-Plantar Erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 0 | 0 | 3 | 1
Dermatitis Acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Decubitus Ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hair Colour Changes (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Rash Papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin Discolouration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin Irritation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 5 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 4 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 0 | 2 | 7 | 3
Proteinuria (Renal and urinary disorders) | 1 | 1 | 7 | 0
Dysuria (Renal and urinary disorders) | 0 | 0 | 2 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 2 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 2 | 0
Nocturia (Renal and urinary disorders) | 0 | 0 | 1 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary Retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 4 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Confusional State (Psychiatric disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Hallucination, Auditory (Psychiatric disorders) | 0 | 0 | 1 | 0
Mental Status Changes (Psychiatric disorders) | 0 | 0 | 1 | 0
Panic Attack (Psychiatric disorders) | 0 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Arteriosclerosis Coronary Artery (Cardiac disorders) | 0 | 0 | 1 | 0
Bradycardia (Cardiac disorders) | 0 | 1 | 0 | 0
Supraventricular Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
Dry Eye (Eye disorders) | 0 | 0 | 1 | 0
Lacrimation Increased (Eye disorders) | 0 | 0 | 1 | 0
Photophobia (Eye disorders) | 0 | 0 | 1 | 0
Strabismus (Eye disorders) | 0 | 1 | 0 | 0
Stoma Site Pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Stoma Site Haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Ear Pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Hearing Impaired (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Malignant Pleural Effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Pelvic Pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Vaginal Haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Allergic Oedema (Immune system disorders) | 0 | 0 | 0 | 1
Stoma Site Infection (Infections and infestations) | 0 | 0 | 1 | 0
Activated Partial Thromboplastin Time Prolonged (Investigations) | 0 | 0 | 1 | 0
Blood Bilirubin Increased (Investigations) | 0 | 0 | 1 | 1
Ejection Fraction Decreased (Investigations) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 3 | 7 | 4
Small Intestinal Obstruction (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Cytomegalovirus Gastrointestinal Infection (Infections and infestations) | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Alanine Aminotransferase Increased (Investigations) | 1 | 0 | 8 | 2

LIMITATIONS AND CAVEATS:
The study was terminated by the sponsor at the end of Phase 1b due to a change in corporate strategy, hence Phase 2 was not carried out.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No